CLINICAL TRIAL: NCT00487123
Title: A Multi-Center, Randomized, Proof-of-Concept, Parallel Control Study With Remind Cap® in Patients With Essential Hypertension and Newly Treated With Valsartan+/-Hydrochlorothiazide (HCTZ)
Brief Title: Efficacy of the New Closure Device in Improving Patient Compliance in Treatment of Hypertension With Valsartan+/-Hydrochlorothiazide (HCTZ) at 6 Months
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVAH631BSG02
Record Dates: First submitted 2007-06-13; First posted 2007-06-15 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Hypertension
Keywords: Hypertension, compliance, Valsartan, hydrochlorothiazide (HCTZ)
MeSH Terms: conditions — Hypertension; Patient Compliance

INTERVENTIONS:
Drug: Valsartan+/- Hydrochlorothiazide

SUMMARY:
This study will evaluate the efficacy of the reminder device Remind Cap® in improving patients' compliance in the consumption of Valsartan +/- Hydrochlorothiazide (HCTZ) in the treatment of hypertension

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypertension that have newly started using Valsartan+/-HCTZ

Exclusion Criteria:

* Pregnancy or Hypersensitivity to Valsartan+/-HCTZ

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Compliance rate at month 3, 6 and post study month 1 will be assessed by pill count

SECONDARY OUTCOMES:
Patient Adherence to study/follow up visits -Clinical Outcome Measurement: Mean sitting systolic BP and mean sitting diastolic BP -Patient's and Physician's Satisfaction Survey

CONTACTS AND LOCATIONS:
Overall Officials: non IND, Study Chair — Sponsor GmbH
Locations (1):
- Novartis Investigative Site, Singapore, Singapore